CLINICAL TRIAL: NCT03827772
Title: Fecal Microbiota Transplantation in Severe Alcoholic Hepatitis- Assessment of Impact on Prognosis and Short-term Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor and Head, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGIMER Hepatology
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Fecal microbiota transplantation (Experimental): 30 grams of stool homogenized with 100 mL of normal saline administered a single time via nasojejunal tube.
  Interventions: Other: Fecal Microbiota Transplantation
- Control Arm (Other): Nutritional supplementation, supportive management
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — 30 grams of stool homogenized with 100 mL of normal saline administered a single time via nasojejunal tube.
  Arms: Intervention Arm: Fecal microbiota transplantation
Other: Standard of care treatment — Nutritional supplementation, supportive management.
  Arms: Control Arm

SUMMARY:
Alcoholic liver disease has become one of the foremost causes of chronic liver disease across the world, and a cause of considerable morbidity and mortality. Alcoholic steatohepatitis is an entity in this broad spectrum, with severe alcoholic hepatitis transitioning to acute on chronic liver failure carrying a one month mortality of as high as 20 to 50%.

The current management guidelines for severe alcoholic hepatitis show benefit with prolonged alcohol abstinence, nutritional support, the use of corticosteroids, pentoxifylline or N-acetyl cysteine (NAC) and early liver transplantation. However, major studies and meta-analyses have demonstrated that these interventions, with the exception of early liver transplantation, do not improve mortality rates to the level of statistical significance. Owing to the high short term mortality associated with severe alcoholic hepatitis, the inadequacy of a treatment that could significantly impact this short term mortality, and the limited applicability of early liver transplantation, a study on newer modalities of treatment is warranted.

The role that human gut microbiota plays in health and disease is receiving considerable attention. Targeting intestinal dysbiosis, a phenomenon found to be intricately linked with the causation of alcoholic hepatitis, could provide insights into novel therapeutic strategies.

Fecal microbiota transplantation is a novel approach that has gained widespread acceptance in in the management of recurrent severe Clostridium difficile infection. It's role is also being studied in other diseases where an association with gut dysbiosis has been found, such as in inflammatory bowel disease and irritable bowel syndrome. The role of FMT has also been studied in liver diseases such as non-alcoholic fatty liver disease (NAFLD), liver cirrhosis and primary sclerosing cholangitis. In this process, a diseased recipient is transferred fecal material containing the microflora of a healthy individual. It limits the colonization of pathogens, inducing colonization resistance, affects microbiota composition in the gut, as well as metabolism in the microbial pathogens. FMT helps alleviate gut dysbiosis and restores gut microbial diversity.

Our aim is to evaluate the role of FMT on short term survival and improvement in scores of prognostic significance (CTP, MELD, MELDNa, mDF) in patients with severe alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Severe alcoholic hepatitis will be defined as proposed by the American College of Gastroenterology

  1. Rapid development or worsening of jaundice and liver-related complications with serum total bilirubin more than 3 milligrams per decilitre.
  2. Aspartate aminotransferase and alanine aminotransferase elevated to more than one and half times the upper limit of normal, but less than 400 IU per litre, with AST to ALT ratio over 1.5.
  3. Documentation of persistent heavy alcohol use until 8 weeks before onset of symptoms.
  4. Alcohol Consumption in female over 40 grams per day for at least 6 months and in males over 60 grams per day for at least 6 months.
  5. Maddrey's Discriminant Function Score of more than 32 OR
  6. A patient of alcoholic hepatitis who will present with grade 1 or 2 of hepatic encephalopathy.

Exclusion Criteria:

1. Intestinal paralysis, lack of bowel sounds, intestinal perforation.
2. Uncontrolled infections.
3. Uncontrolled upper gastrointestinal bleeding.
4. Grade 3,4 hepatic encephalopathy.
5. Hepatic or extrahepatic malignancy.
6. Maddrey's Discriminant Function (mDF) >90 or MELD>30.
7. Autoimmune hepatitis, Wilson's disease, suspected drug induced liver injury.
8. Patients who are aged >60 years
9. WBC count <1000 cells/mm3
10. Pregnancy or nursing.
11. Human Immunodeficiency Virus (HIV), HBV, HCV infection.
12. Patient's unwillingness to participate in the study.
13. Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 months

SECONDARY OUTCOMES:
Improvement in CTP (Child Turcotte Pugh Score) | 3 months
Improvement in MELD score | 3 months
Improvement in MELDNa score | 3 months
Improvement in CLIF SOFA score | 3 months
Improvement in mDF | 3 months
Changes in inflammatory markers (IL1b, IL6, TNF α) pre and post FMT, | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma A, Roy A, Premkumar M, Verma N, Duseja A, Taneja S, Grover S, Chopra M, Dhiman RK. Fecal microbiota transplantation in alcohol-associated acute-on-chronic liver failure: an open-label clinical trial. Hepatol Int. 2022 Apr;16(2):433-446. doi: 10.1007/s12072-022-10312-z. Epub 2022 Mar 28. PMID 35349076